CLINICAL TRIAL: NCT03453463
Title: Impact of Exercise on Sarco-osteopenia in Community Dwelling Men 70 Years and Older. A Randomized Controlled Trial
Brief Title: Exercise Effects on Sarco-Osteopenia in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FROST
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia; Osteopenia
Keywords: sarcopenia; osteopenia; older men; community dwelling; physical functioning
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor are not aware of participant status and are nor allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise and protein supplementation (Experimental): Predominately resistance exercise training 2-3x week for 18 months; 1.5-1.7 g/kg/d total protein supplementation, Calcium and Vitamin-D-supplementation (i.e. 800 mg/800 IE/d)
  Interventions: Other: exercise
- control (No Intervention): Calcium and Vitamin-D-supplementation (i.e. 800 mg/800 IE/d)

INTERVENTIONS:
Other: exercise — 3x week predominately resistance exercise for 18 months
  Other Names: resistance exercise
  Arms: exercise and protein supplementation

SUMMARY:
The study determined the effects of predominately resistance type exercise in combination with protein supplements on parameters of sarcopenia and osteopenia (sarco-osteopenia) in older, community dwelling men with sarcopenia and -osteopenia over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenia according to Baumgartner et al.(SMI: > -2 SD* T-Score)
* Osteopenia at the lumbar spine or hip according to WHO (> -1 SD T-Score)
* community dwelling people
* able to transfer to our lab

Exclusion Criteria:

* secondary osteoporosis
* history of hip fracture
* medication/diseases that relevantly affect muscle/bone metabolism (last 2 years)
* alcohol abuses of more than 60 g/d ethanol
* cardio-vascular diseases that prevent exercise
* very low physical capacity that prevent exercise in a group setting

SD: Standard Deviation

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Lumbar spine Bone Mineral Density (QCT) | changes from baseline to 18 months
  Lumbar spine Bone Mineral Density as determined by Quantitative Computed Tomography

SECONDARY OUTCOMES:
Lumbar spine Bone Mineral Density (DXA) | changes from baseline to 12 and 18 months
  Lumbar spine Bone Mineral Density as determined by dual-energy x-ray absorptiometry (DXA)
Femoral Neck Bone Mineral Density | changes from baseline to 12 and 18 months
  Total hip Bone Mineral Density as determined by dual-energy x-ray absorptiometry (DXA)
Skeletal muscle mass index | changes from baseline to 6, 12 and 18 months
  Skeletal muscle mass as defined fat and bone free mass of the limbs as determined by DXA divided by square height
Gait velocity | changes from baseline to 6, 12 and 18 months
  Habitual gait speed over 10 m
Hand-grip strength | changes from baseline to 6, 12 and 18 months
  Maximum hand-grip strength of the dominant and non-dominant hand as assessed by a Jamar dynamometer
Hip and leg extensor strength | changes from baseline to 6, 12 and 18 months
  Maximum dynamic hip and leg extensor strength as determined by a isokinetic leg press
Muscle Density at the calf, thigh and para-vertebral site | changes from baseline to 6 and 12 months
  Muscle Density at the calf, thigh and para-vertebral site as assessed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Engelke, PhD, Study Chair — Institute of Medical Physics, University of Erlangen-Nürnberg, Germany
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nürnberg, Germany, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kemmler W, Bebenek M, Kohl M, von Stengel S. Exercise and fractures in postmenopausal women. Final results of the controlled Erlangen Fitness and Osteoporosis Prevention Study (EFOPS). Osteoporos Int. 2015 Oct;26(10):2491-9. doi: 10.1007/s00198-015-3165-3. Epub 2015 May 12. PMID 25963237
- [Background] Kemmler W, von Stengel S. Bone: High-intensity exercise to prevent fractures - risk or gain? Nat Rev Endocrinol. 2018 Jan;14(1):6-8. doi: 10.1038/nrendo.2017.148. Epub 2017 Nov 10. No abstract available. PMID 29125144
- [Background] Kemmler W, von Stengel S, Kohl M. Exercise frequency and bone mineral density development in exercising postmenopausal osteopenic women. Is there a critical dose of exercise for affecting bone? Results of the Erlangen Fitness and Osteoporosis Prevention Study. Bone. 2016 Aug;89:1-6. doi: 10.1016/j.bone.2016.04.019. Epub 2016 Apr 21. PMID 27108341
- [Derived] Kircher K, Chaudry O, Nagel AM, Ghasemikaram M, Uder M, Jakob F, Kohl M, Kemmler W, Engelke K. Effects of high-intensity training on fatty infiltration in paraspinal muscles in elderly males with osteosarcopenia - the randomized controlled FrOST study. BMC Geriatr. 2024 Feb 8;24(1):141. doi: 10.1186/s12877-024-04736-5. PMID 38326734
- [Derived] Kemmler W, Kohl M, von Stengel S, Schoene D. Effect of high-intensity resistance exercise on cardiometabolic health in older men with osteosarcopenia: the randomised controlled Franconian Osteopenia and Sarcopenia Trial (FrOST). BMJ Open Sport Exerc Med. 2020 Dec 24;6(1):e000846. doi: 10.1136/bmjsem-2020-000846. eCollection 2020. PMID 33408874
- [Derived] Kemmler W, Kohl M, Frohlich M, Schoene D, von Stengel S. Detraining effects after 18 months of high intensity resistance training on osteosarcopenia in older men-Six-month follow-up of the randomized controlled Franconian Osteopenia and Sarcopenia Trial (FrOST). Bone. 2021 Jan;142:115772. doi: 10.1016/j.bone.2020.115772. Epub 2020 Nov 26. PMID 33249320